CLINICAL TRIAL: NCT01367899
Title: Conserve Plus Total Hip Resurfacing System: A Non-Randomized, Multi-center, NewEnrollement Post Approval Study
Brief Title: CONSERVE Plus Post-Approval Study (PAS)
Status: Terminated | Type: Observational
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 09-LJH-002
Record Dates: First submitted 2011-05-02; First posted 2011-06-07 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Other and Unspecified Injury to Hip and Thigh
Keywords: Safety; Efficacy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CONSERVE® Plus hip resurfacing: Recipients/C Plus (IDE)study

SUMMARY:
The objective of this post-approval study is to provide scientifically valid and reliable evidence that supports claims of longer term safety and effectiveness with regard to Month 120 device survivorship rates.

DETAILED DESCRIPTION:
This study will evaluate the performance of CONSERVE Plus Hip Resurfacing System under actual conditions of use. Additionally, this study will evaluate the performance of the device in the post approval environment to see if there are any significant changes in device performance as compared to the pre-market IDE Study

ELIGIBILITY:
Inclusion Criteria:

1. Was previously enrolled in the CONSERVE® Plus IDE as part of the All Enrolled Audited Cohort (N=1366 procedures (1206 patients)) and received the "Original Shell".
2. Is willing and able to comply with the study plan and able to understand and sign the Patient Informed Consent Form.

Exclusion Criteria:

1. Patient is mentally incompetent.
2. Patient is a prisoner.
3. Patient is an alcohol and/or drug abuser
4. Patient has undergone device revision or removal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have already undergone hip resurfacing in the CONSERVE Plus IDE.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2010-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Clinical success at Month 120 | 10 years
  Clinical success at Month 120 for each patient will be survivorship, defined as freedom from revision or removal for any aseptic reason and at least "good" function/pain relief defined as Harris Hip Score ≥ 80.

SECONDARY OUTCOMES:
Radiographic outcomes | 10 years
  Secondary measures: radiographic outcomes
Metal Ion (serum) | 24 months
  metal ion (serum) and renal function will also be collected.
Assessment for Adverse Events | 10 years
  Subjects will be assessed for any adverse events during their length of participation
Measurement of Patient Satisfaction | 10 years
  Patient satisfaction as assessed by the SF-12

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bolognesi, MD, Principal Investigator — Duke University
Locations (1):
- Michael Bolognesi, MD, Durham, North Carolina, United States